CLINICAL TRIAL: NCT06030375
Title: Safety, Tolerability and Pharmacokinetics After Continuous Infusion of KAND567. A Single-centre, Placebo-controlled, Randomised, Double-blind Study in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics After Continuous Infusion of KAND567
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novakand Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KAN0004; 2019-004585-18 (EudraCT Number)
Record Dates: First submitted 2023-08-24; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The physical appearance of the KAND567 solution is a clear transparent solution with a distinct smell. An unblinded pharmacist or registered nurse at the study centre therefore prepared the dosing solutions.
  There were two unblinded persons working together, one person handled the IMP and perform the dispensing according to the randomisation list and the other person monitored the process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KAND567 in ascending doses (Active Comparator): In each of the 3 cohorts, 6 subjects were planned to be randomised to receive KAND567. The dose levels were 33.8 mg/6 h (cohort 1), 67 mg/6 h (cohort 2), or 134 mg/6 h (cohort 3).
  Interventions: Drug: KAND567
- Placebo (Placebo Comparator): In each of the 3 cohorts, 2 subjects were planned to be randomised to receive Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KAND567 — Continuous intravenous infusion for 6 hours
  Arms: KAND567 in ascending doses
Other: Placebo — Continuous intravenous infusion for 6 hours
  Arms: Placebo

SUMMARY:
The study was planned to consist of 24 healthy subjects in 3 dosing cohorts receiving a continuous i.v. infusion of KAND567 or placebo for 6 h (6 subjects on active and 2 subjects on placebo per cohort), with the option of two additional cohorts of the same size and group composition.

DETAILED DESCRIPTION:
The 3 planned dose levels of KAND567 were based on preliminary data from previous i.v. infusions and were chosen to obtain approximate Css levels of 0.5, 1.0 and 2.0 μM. The dose levels were 33.8 mg/6 h (cohort 1), 67 mg/6 h (cohort 2), or 134 mg/6 h (cohort 3).

Each cohort of participants was planned to consist of 8 subjects (2 on placebo and 6 on active drug), i.e. a total of 24 subjects. A sentinel approach was used for all three cohorts, starting dosing with two subjects (one on active drug, one on placebo). If safe and tolerable, an additional two or three subjects will be administered. If safe and tolerable, the remaining three or four subjects of the cohort were dosed. There was an evaluation of safety and tolerability from the previous cohort prior to proceeding to the next cohort.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study specific procedures
* Body weight > 50 kg
* Body Mass Index (BMI) ≥ 19 and ≤ 30 kg/m^2 at screening
* Healthy male and female subjects aged ≥ 18 and ≤ 65 years at screening
* Male subjects must agree to use an adequate method of contraception. Male subjects who are heterosexually active must use, with their partner, a condom AND one of the following methods of highly effective contraception from the time of IMP administration until 90 days after dosing of IMP.

  * oral (except low-dose gestagen (lynestrenol and norestisteron)), injectable or implanted hormonal contraceptives
  * intrauterine device
  * intrauterine system (for example progestin-releasing coil)
  * vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate)
  * bilateral tubal occlusion or hysterectomy
* Female subject must be of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy or bilateral oophorectomy; or as post-menopausal females defined as 12 months' amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulating hormone 25-140 IE/L and estradiol < 200 pmol/L is confirmatory])
* Willingness and ability to comply with study procedures, visit schedules, study restrictions and requirements

Exclusion Criteria:

* Present or known history of clinically significant cardio- or cerebrovascular, pulmonary, renal, hepatic, neurological, mental, metabolic, endocrine, haematological, gastrointestinal disorder, significant respiratory disease, sleep apnoea, narcolepsy or any other major disorder that may interfere with the objectives of the study, as judged by the investigator
* Any clinically significant abnormalities in physical examination, electrocardiogram (ECG; e.g. QTcF>450 ms), clinical chemistry, haematology or urinalysis results at screening, as judged by the investigator
* Clinically significant abnormal blood pressure (treated or untreated), defined as systolic pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 90 mmHg at screening
* Pulse rate < 45 bpm at screening
* Clinically significant illness within the 5 days prior to the administration of the IMP
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody or human immunodeficiency virus (HIV)
* Known or suspected drug or alcohol abuse or positive screen for drugs of abuse test or positive alcohol breath test at screening visit or any time prior to randomisation
* Smoking > 5 cigarettes per day, or inability to refrain from smoking or using other nicotine-containing products during the stay at the study centre.
* Subject who has received any investigational drug within the last 3 months before administration of IMP
* Plasma donation within one month of screening visit, or any blood donation/ blood loss > 450 mL during the 3 months prior to screening visit
* Use of the herbal remedy St. John's Wort within two weeks prior to the first dose of the IMP (induces cytochrome P450-3A4)
* Use of prescribed medication during the two weeks prior to the administration of the IMP (or longer if the prescribed medication has a half-life long enough to potentially expose the subject to any significant systemic exposure, as judged by the investigator)
* Use of over-the-counter drugs (including herbals (St. John's Wort - see above), vitamins and minerals) during one week prior to the administration of the IMP or need for concomitant medication during the study. However, occasional paracetamol for pain relief is allowed (up to 3 g per 24 hours)
* Female subjects: Positive pregnancy test at screening visit or at any time prior to randomisation
* Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements
* Subject has an eGFR < 80 mL/min/1.73m^2 at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability after continuous infusion of KAND567, as measured by adverse events (AEs) | From the first IMP administration (Day 1) until the last follow-up visit (Day 30)
  Measured by the occurrence of AEs and serious adverse events (SAEs)
Safety and tolerability after continuous infusion of KAND567, as measured by vital signs | From the first IMP administration (Day 1) until the last follow-up visit (Day 30)
  Measured by the occurrence of clinically abnormal vital signs
Safety and tolerability after continuous infusion of KAND567, as measured by ECG | From the first IMP administration (Day 1) until the last follow-up visit (Day 30)
  Measured by the occurrence of clinically abnormal electrocardiography (ECG)
Safety and tolerability after continuous infusion of KAND567, as measured by lab safety tests | From the first IMP administration (Day 1) until the last follow-up visit (Day 30)
  Measured by the occurrence of clinically abnormal lab test results (routine clinical chemistry, haematology, and urinalysis)
Pharmacokinetics (PK) after continuous infusion of KAND567, as measured by Css | From the first IMP administration (Day 1) until Day 2
  Measured by plasma drug concentration at steady state (Css)
Pharmacokinetics (PK) after continuous infusion of KAND567, as measured by AUC | From the first IMP administration (Day 1) until Day 2
  Measured by the area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) after continuous infusion of KAND567, as measured by t1/2z | From the first IMP administration (Day 1) until Day 2
  Measured by terminal half-life (t1/2z)
Pharmacokinetics (PK) after continuous infusion of KAND567, as measured by Vss | From the first IMP administration (Day 1) until Day 2
  Measured by the apparent volume of distribution at steady state (Vss)
Pharmacokinetics (PK) after continuous infusion of KAND567, as measured by CL | From the first IMP administration (Day 1) until Day 2
  Measured by the systemic clearance (CL)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, PhD, Principal Investigator — Clinical Research Services Turku (CRST)
Locations (1):
- Clinical Research Services Turku (CRST), Turku, Finland

IPD SHARING:
Plan to Share IPD: No